CLINICAL TRIAL: NCT04806464
Title: A Dose Ascending, Open Phase I Clinical Study to Evaluate the Safety, Tolerability , Pharmacokinetics Characteristics and Preliminary Effectiveness of VG161 in Subjects with Advanced Primary Liver Cancer
Brief Title: Clinical Study of VG161 in Subjects with Advanced Primary Liver Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CNBG-Virogin Biotech (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-C102
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Liver Cancer
Keywords: Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VG161 (Experimental): Part1:
  1. 1.0*10^8 PFU on Day 1(1.0×10^8PFU)
  2. 1.0*10^8 PFU on Days 1 to 2(2.0×10^8PFU)
  3. 1.0*10^8 PFU on Days 1 to 3(3.0×10^8PFU)
  4. 1.3*10^8 PFU on Days 1 to 3(4.0×10^8PFU)
  5. 1.7*10^8 PFU on Days 1 to 3(5.0×10^8PFU)
  Part2:
  Depends on the recommended dose in Part1
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell))

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) — Intratumoral injection only. The dosing date can be the Day 1 only or Days 1 through 5.
  Other Names: VG161

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 Injectable. This phase I study will be conducted in HSV-seropositive subjects with advanced primary liver cancer that are refractory to conventional therapies. This is an open label study and it's divided into two parts.

Part 1: This part is ascending dose design to determine the safety and tolerability of VG161 and find recommended dose of VG161.

Part 2: This part is extended dose design to determine the effectiveness of VG161.

DETAILED DESCRIPTION:
Part 1: This part will be conducted in 5 dose ascending cohorts, including 2 accelerated titration design dose group and 3 dose escalation groups. Descriptive statistics will be used to summarize data.

Part 2: This part will only include the part 1 recommended dose. Hypothesis test and descriptive statistics will be used to summarize data.

ELIGIBILITY:
1. According to 'The Diagnostic and Therapeutic Criteria for Primary Liver Cancer' (NMPA, 2019 Edition), subject with advanced primary hepatocellular carcinoma, intrahepatic cholangiocarcinoma, combined hepatocellular which is refractory/relapsed after and/or intolerant of standard therapies or for which no standard therapy exists. For the second stage of Simon's two-stage in part 2, only patients with advanced primary hepatocellular carcinoma will be enrolled.
2. There are tumor lesions intrahepatic and / or extrahepatic metastases that can be injected under B ultrasound and meet the volume requirements of the current dose group, and the longest diameter of injectable tumor lesion >1.5cm（or the shortest diameter of lymph node lesions）
3. Eastern Cooperative Oncology Group (ECOG) scores 0 or 1.
4. Life expectancy is at least 3 months.
5. Required organ function:

1) Hematology blood (no blood transfusion or colony stimulating factor treatment within 14 days): absolute neutrophil count (ANC)≥1.5×10^9L, platelets (PLT)≥75×10^9L, hemoglobin (Hb)≥85g/L; 2) Liver function: Total Serum bilirubin (TBIL)≤1.5×ULN (the upper limit of the reference range), Alanine aminotransferase (ALT)≤5×ULN, aspartate aminotransferase (AST)≤5×ULN; 3)Child-Pugh A-B level; 4) Renal function: Serum creatinine≤1.5×ULN, and creatinine clearance≥45 ml/min (calculated per Cockcroft-Gault formula); 5) Coagulation function: activated partial thromboplastin time (APTT)≤1.5×ULN, prothrombin time(PT) ≤1.5×ULN, international standardized ratio (INR)≤1.5×ULN.

6. Subjects who are HBV-DNA negative; or HBV-DNA positive are required to receive treatment in accordance with the 'Guidelines for the prevention and treatment of chronic hepatitis B' (2019 Edition) or clinical practice.

7.Subjects of childbearing potential (male and female) must agree to use a reliable contraceptive method (hormone or barrier method or abstinence) during the study and for at least 90 days following the last dose; females of childbearing potential must have a negative blood pregnancy test within 7 days of study enrollment.

8.Signed written informed consent.

Exclusion Criteria:

1. Subject in prior anti-tumor therapies such as chemotherapy, radiotherapy, biotherapy, endocrinotherapy, targeted therapy, immunotherapy within 4 weeks of study treatment initiation. Oral fluorouracil analogues and small molecule targeted drugs were 2 weeks prior to the first dose of study drug or within 5 half-lives of the drug (whichever was longer).
2. Transcatheter arterial chemoembolization(TACE) within 4 weeks of study treatment initiation
3. Participation in clinical trials of any other investigational agents within 4 weeks of study treatment initiation.
4. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks of study treatment initiation.
5. Patients who received systemic treatment with either corticosteroids ( >10 mg/ daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study treatment initiation.
6. Subjects with any ≥Grade 1 toxicity (as per NCI CTC AE Version 5.0) related to prior anti-cancer therapy (except for toxicity that the investigator assessed to be no safety risk, such as alopecia.).
7. Subjects with Central Nervous System (CNS) metastasis or meningeal metastasis .
8. Seronegative for Herpes Simplex Virus (HSV) (HSV-1IgG and HSV-1IgM).
9. Subjects with the relapse of HSV infection and relevant clinical manifestations, such as lip herpes, herpes keratitis, herpes dermatitis, and genital herpes.
10. Subjects with other uncontrolled active infections.
11. Known history of immunodeficiency and test positive of human immunodeficiency virus (HIV).
12. History of severe cardiovascular disease:

1)Ventricular arrhythmias requiring clinical intervention; 2)QTc interval >480 ms; 3)Acute coronary syndrome, congestive heart failure, stroke or other cardiovascular events of III grade or above within 6 months; 4)The cardiac function grade≥II or left ventricular ejection fraction (LVEF) <50% per the New York Heart Association (NYA); 5)Uncontrolled hypertension.

13. Subjects with active or past autoimmune diseases that are likely to recur (e.g. systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.); acceptable for patients with clinically stable autoimmune thyroiditis.

14. Previous immunotherapy with an immune-related adverse event (irAE) such as immune-related pneumonia, myocarditis, etc., which, in the judgement of the investigator, may affect the safety of the investigational drug. 15. known to have alcohol or drug dependence. 16. Persons with mental disorders or poor compliance. 17. Pregnant or lactating women. 18. Subjects with any significant unrelated systemic illness that to the investigator's opinion would compromise the subject's eligibility to participate the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Part1: MTD/Recommended dose | 7 month
  MTD (Maximum tolerable dose) /Recommended dose
Part1: Occurence of DLT | 1month
  Occurence of DLT (Dose Limiting Toxicity)
Part1: Numbers of DLT | 1 month
  Numbers of DLT (Dose Limiting Toxicity)
Part1: Occurence of AE and SAE（NCI CTCAE 5.0） | 7 months
  Occurence of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part1: Frequency of AE and SAE（NCI CTCAE 5.0） | 7 months
  Frequency of Adverse Event (AE) and Serious Adverse Event (SAE) （NCI CTCAE 5.0）
Part2:ORR | 7 months
  Evaluate Objective Response Rate by RECIST 1.1

SECONDARY OUTCOMES:
Part1:Tmax(h) | At the end of Cycle 1 (each cycle is 28 days)
  Time to peak
Part1:Cmax(copies/ugDNA) | At the end of Cycle 1 (each cycle is 28 days)
  Maximum concentration
Part1:ORR | 7 months
  Evaluate Objective Response Rate by iRECIST
Part1:DOR | 7 months
  Evaluate Disease Control Rate by iRECIST
Part1:PFS | 7 months
  Evaluate medium Progression Free Survival by iRECIST
Part1:OS rate | 17 months
  Evaluate Overall Survival rate
Part 1:CD3+, CD4+, CD8+ | 7 months
  Concentration of CD3+, CD4+, CD8+
Part 1:IL15 | 7 months
  Concentration of IL15
Part 1:PD-L1, PD-1 | 7 months
  Concentration of PD-L1, PD-1
Part 2:PFS | 7 months
  Evaluate medium Progression Free Survival by iRECIST
Part 2:OS rate | 17 months
  Evaluate Overall Survival rate
Part 2: OS | 17 months
  Overall Survival
Part 2:DOR | 7 months
  Evaluate Disease Control Rate by iRECIST
Part 2:Safety indicators：AEs | 7 months
  Incidence of adverse events (NCI CTCAE 5.0)
Part 2:Safety indicators：ECOG | 7 months
  Incidence of abnormal ECOG scores
Part 2:Safety indicators：12-lead electrocardiograms | 7 months
  Incidence of abnormal 12-lead electrocardiograms
Part 2:Safety indicators：laboratory tests results | 7 months
  Incidence of abnormal laboratory tests results
Part 2:CD3+, CD4+, CD8+ | 7 months
  Concentration of CD3+, CD4+, CD8+
Part 2:IL15 | 7 months
  Concentration of IL15
Part 2:PD-L1, PD-1 | 7 months
  Concentration of PD-L1, PD-1

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen Y, Bai X, Zhang Q, Liang X, Jin X, Zhao Z, Song W, Tan Q, Zhao R, Jia W, Gu S, Shi G, Zheng Z, Wei G, Wang Y, Fang T, Li Y, Wang Z, Yang Z, Guo S, Lin D, Wei F, Wang L, Sun X, Qin A, Xie L, Qiu Y, Bao W, Rahimian S, Singh M, Murad Y, Shang J, Chu M, Huang M, Ding J, Chen W, Ye Y, Chen Y, Li X, Liang T. Oncolytic virus VG161 in refractory hepatocellular carcinoma. Nature. 2025 May;641(8062):503-511. doi: 10.1038/s41586-025-08717-5. Epub 2025 Mar 19. PMID 40108464